CLINICAL TRIAL: NCT02673983
Title: Endoscopic Full-thickness Biopsy of the Intestine
Brief Title: Safety and Efficacy Study of the FTRD System for Obtaining Full-thickness Intestinal Biopsies
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was never started
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EFAT-001
Record Dates: First submitted 2016-01-15; First posted 2016-02-04 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Gastrointestinal Motility Disorders
Keywords: Intestinal; Biopsy; full thickness; endoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients undergoing endoscopic full-thickness biopsy (Experimental)
  Interventions: Procedure: Endoscopic full-thickness biopsy

INTERVENTIONS:
Procedure: Endoscopic full-thickness biopsy

SUMMARY:
The aim of this study is to evaluate FTRD (full-thickness resection device) in terms of obtaining full-thickness biopsies form the gastrointestinal tract endoscopically in the work-up of patients with gastrointestinal motility disorders.

DETAILED DESCRIPTION:
Functional intestinal disorders are a common problem and diagnosis is a challenge to clinicians. Several motility disorders are caused by pathological changes in the neuromuscular network in the intestinal wall. To obtain a diagnosis a full-thickness biopsy is required. At present, this kind of biopsy is usually obtained by a laparoscopic surgical procedure, requiring full anesthesia, operating room and several days of postoperative care in the hospital. Today, there is lacking a more minimal invasive approach for obtaining full-thickness biopsies from the gastrointestinal tract. A new device has been developed called full-thickness resection device (FTRD), which has proved useful and safe from removing polyps in the gastrointestinal tract (Schmidt A Endoscopy 47;8, 719-725). The specific aims of this study is to determine if FTRD safe for obtaining full-thickness biopsies form the gastrointestinal tract and whether these FTRD biopsies be used for clinical diagnosis of patients with suspected intestinal motility disorders. If these aims can be achieved FTRD would be of potential great value for patients and health care in the management of patients with gastrointestinal disorders. 40 patients will be included, i.e. 10 patients will undergo FTRD biopsy in the sigmoid colon, distal ileum, jejunum and duodenum. Patients will undergo the biopsy procedure under conscious sedation at the Endoscopy Unit in Malmö, Region Skane and stay one night at the hospital to detect any complications. A venous blood sample will be taken before and 24 hours after the biopsy for examination of systemic inflammatory changes. All biopsies will examined by an expert in neuromuscular pathology.

ELIGIBILITY:
Inclusion Criteria:

* Patients with functional gastrointestinal motility disorders in which a full-thickness biopsy is needed to obtain a clinical diagnosis.

Exclusion Criteria:

* Patients less than 18 years old and patients not giving consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Safety: The number of patients with bleeding or perforation will be determined and reported. | 24 hours
  Upon signs of clinical significant bleeding a colonoscopy will be performed and upon clinical signs of perforation will the patient undergo a computer tomography. The number of patients with bleeding or perforation will be determined and reported.

SECONDARY OUTCOMES:
Efficacy: The number of patients in which a clinical diagnosis was obtained based on the full thickness biopsy will be determined and reported. | 4-8 weeks when pathological examination is completed
  The number of patients in which a clinical diagnosis was obtained based on the full thickness biopsy will be determined and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Thorlacius, MD, PhD, Principal Investigator — Region Skane, Department of Surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schmidt A, Bauerfeind P, Gubler C, Damm M, Bauder M, Caca K. Endoscopic full-thickness resection in the colorectum with a novel over-the-scope device: first experience. Endoscopy. 2015 Aug;47(8):719-25. doi: 10.1055/s-0034-1391781. Epub 2015 Mar 12. PMID 25763833